CLINICAL TRIAL: NCT00836004
Title: Randomized, 2-Way Crossover, Bioequivalence Study of Clindamycin 300 mg Capsules and Cleocin Hcl Administered as 1 x 300 mg Capsule in Healthy Subjects Under Fed Conditions
Brief Title: Clindamycin 300 mg Capsules in Healthy Subjects Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 30313
Record Dates: First submitted 2009-02-03; First posted 2009-02-04 (Estimated); Results first posted 2009-07-21 (Estimated); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Healthy
Keywords: Bioequivalence; Healthy Subjects
MeSH Terms: interventions — Clindamycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clindamycin (test) (Experimental): Clindamycin 300 mg Capsule (test) dosed in first period followed by Cleocin® 300 mg Capsule (reference) dosed in second period
  Interventions: Drug: Clindamycin 300 mg capsule
- Cleocin® (reference) (Active Comparator): Cleocin® 300 mg Capsule (reference) dosed in first period followed by Clindamycin 300 mg Capsule (test) dosed in second period
  Interventions: Drug: Cleocin HCl 300 mg capsules

INTERVENTIONS:
Drug: Clindamycin 300 mg capsule — 1 x 300 mg
  Arms: Clindamycin (test)
Drug: Cleocin HCl 300 mg capsules — 1 x 300 mg
  Arms: Cleocin® (reference)

SUMMARY:
The objective of this study is to compare the rate and extent of absorption of clindamycin 300 mg capsules (test) versus Cleocin HCl (reference, administered as 1 x 300 mg capsule under fed conditions.

DETAILED DESCRIPTION:
Criteria for Evaluation: FDA Bioequivalence Criteria

Statistical Methods: FDA bioequivalence statistical methods

ELIGIBILITY:
Inclusion Criteria:

* Child-bearing potential or non-child-bearing potential female or male, non-smoker, ≥ 18 and ≤65 years of age.
* Non-child-bearing potential female subject is defined as follows:

  1. Post-menopausal state: absence of menses for 12 months prior to drug administration or hysterectomy with bilateral oophorectomy at least 6 months prior to drug administration.
  2. Surgically sterile: hysterectomy, bilateral oophorectomy, or tubal ligation at least 6 months prior to drug administration.
* Capable of consent.

Exclusion Criteria:

* Clinically significant illnesses within 4 weeks prior to the administration of the study medication.
* Clinically significant surgery within 4 weeks prior to the administration of the study medication.
* Any clinically significant abnormality found during the medical screening.
* Any reason which, in the opinion of the Medical Sub-Investigator, would prevent the subject from participating in the study.
* Abnormal laboratory tests judged clinically significant.
* Positive testing for hepatitis B, hepatitis C, or HIV at screening.
* EGC abnormalities (clinically significant) or vital sign abnormalities(systolic blood pressure lower than 90 over 140 mmHg, diastolic blood pressure lower than 50 or over 90 mmHg, or heart rate less than 50 or over 100 bpm) at screening.
* BMI≥ 30.0kg/m2.
* History of significant alcohol abuse within six months prior to the screening visit or any indication of the regular use of more than fourteen units of alcohol per week ( 1 Unit= 150 mL of wine, 360 mL of beer, or 45 mL of 40% alcohol) or positive alcohol breath test at screening.
* History of drug abuse or use of illegal drugs: use of soft drugs (such as marijuana) within 3 months prior to the screening visit or hard drugs (such as cocaine, phencyclidine [PCP] and crack) within 1 year prior to the screening visit or positive urine drug screen at screening.
* History of allergic reactions to clindamycin or other related drugs (e.g. lienomycin).
* History of allergic reactions to heparin.
* Use of any drugs known to induce or inhibit hepatic drug metabolism (examples of inducers: barbiturates, carbamazepine, phenytoin, glucocorticoids, rifampin/rifabutin; examples of inhibitors: antidepressants, cimetidine, diltiazem, erythromycin, ketoconazole, MAO inhibitors, neuroleptics, verapamil, quinidine) within 30 days prior to administration of the study medication.

Use of an investigational drug or participation in an investigational study within 30 days prior to administration of the study medication.

* Clinically significant history or presence of any clinically significant gastrointestinal pathology (e.g. chronic diarrhea, inflammatory bowel diseases), unresolved gastrointestinal symptoms (e.g. diarrhea, vomiting), liver or kidney disease, or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of the drug.
* Any clinically significant history or presence of clinically significant neurological, endocrinal, cardiovascular, pulmonary, haematologic, immunologic, psychiatric, or metabolic disease.
* Use of prescription medication within 14 days prior to administration of study medication or over-the-counter products ( including natural food supplements, vitamins, garlic as supplement) within 7 days prior to administration of study medication, except for topical products without systemic absorption.
* Difficulty to swallow study medication.
* Use of any tobacco products in the 90 days preceding drug administration.
* Any food allergy, intolerance, restriction or special diet that could, in the opinion of the Medical Subinvestigator, contraindicate the subjects's participation in this study.
* A depot injection or an implant of any drug within 3 months prior to administration of study medication.
* Donation of plasma (500 mL) within 7 days prior to drug administration. Donation or loss of whole blood prior to administration of the study medication as follows:

  1. less than 300 mL or whole blood within 30 days,
  2. 300 mL to 500 mL of whole blood within 45 days,
  3. more than 500 mL of whole blood within 56 days prior to drug administration.
* Intolerance to venipunctures.
* Subjects with a clinically significant history of tuberculosis, epilepsy, asthma, diabetes, psychosis, or glaucoma will not be eligible for this study.
* Subjects unable to understand or unwilling to sign the Informed Consent Form.
* Clinically significant history of diarrhea subsequent to administration or antibacterial agents or antibiotics.
* Additional exclusion criteria for females only:

  1. Breast-feeding subject.
  2. Positive urine pregnancy test at screening
  3. Female subjects of childbearing potential having unprotected sexual intercourse with any non-sterile male partner (i.e. male who has not been sterilized by vasectomy for at least 6 months) within 14 says prior to study drug administration. Acceptable methods of contraception:

     1. condom + spermicide,
     2. diaphragm + spermicide,
     3. intra-uterine contraceptive devise (placed at least 4 weeks prior to study drug administration.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2003-11; Primary Completion 2003-11 (Actual); Study Completion 2003-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benoit Girard, M.D., Principal Investigator — Anapharn Inc.
Locations (1):
- Anapharm Inc., Sainte-Foy, Quebec, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Clindamycin (Test) First: Clindamycin 300 mg Capsule (test) dosed in first period followed by Cleocin® 300 mg Capsule (reference) dosed in second period
- Cleocin® (Reference) First: Cleocin® 300 mg Capsule (reference) dosed in first period followed by Clindamycin 300 mg Capsule (test) dosed in second period
Period: First Intervention
Arm/Group | Clindamycin (Test) First | Cleocin® (Reference) First
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0
Period: Washout: 7 Days
Arm/Group | Clindamycin (Test) First | Cleocin® (Reference) First
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Clindamycin (Test) First | Cleocin® (Reference) First
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Clindamycin (Test) First | Cleocin® (Reference) First | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 24
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 5 | 6 | 11
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 12 | 12 | 24
Region of Enrollment [Number; unit: participants]
  Canada | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Cmax - Maximum Observed Concentration
Description: Bioequivalence based on Cmax
Time Frame: Blood samples collected over 24 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Clindamycin: Clindamycin 300 mg Capsule (test) dosed in either period
- Cleocin®: Cleocin® 300 mg Capsule (reference) dosed in either period
Arm/Group | Clindamycin | Cleocin®
Number analyzed (Participants) | 24 | 24
ng/mL | 2936.10 (608.06) | 2955.65 (685.51)
Statistical Analysis 1: Comparison: Clindamycin vs Cleocin®; Test type: Non-Inferiority or Equivalence — Using GLM procedures in SAS, ANOVA (Analysis of Variance) will be performed on log-transformed AUC0-t, AUC0-inf and Cmax at the alpha level of 0.05; Test/Ref Ratio of LS Means x 100 = 99.69, 90% CI [93.88 to 105.85] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

2. Primary Outcome: AUCinf - Area Under the Concentration-time Curve From Time Zero to Infinity (Extrapolated)
Description: Bioequivalence based on AUCinf
Time Frame: Blood samples collected over 24 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Clindamycin | Cleocin®
Number analyzed (Participants) | 24 | 24
ng*h/mL | 14981.11 (4181.02) | 15452.22 (3944.88)
Statistical Analysis 1: Comparison: Clindamycin vs Cleocin®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Test/Ref Ratio of LS Means x 100 = 96.23, 90% CI [90.62 to 102.19] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

3. Primary Outcome: AUC0-t - Area Under the Concentration-time Curve From Time Zero to Time of Last Non-zero Concentration (Per Participant)
Description: Bioequivalence based on AUC0-t
Time Frame: Blood samples collected over 24 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Clindamycin | Cleocin®
Number analyzed (Participants) | 24 | 24
ng*h/mL | 14452.44 (4179.92) | 14761.88 (3894.29)
Statistical Analysis 1: Comparison: Clindamycin vs Cleocin®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Test/Ref Ratio of LS Means x 100 = 97.17, 90% CI [92.14 to 102.48] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prinicipal Investigator is not permitted to discuss or publish trial results.